CLINICAL TRIAL: NCT03260582
Title: Implementation and Assessment of a Life-style Focused Patient Support Application (App) and Activity Trackers for Improving Risk Factor Management, Physical Activity, Quality of Life and Prognosis in Post-myocardial Infarction Patients
Brief Title: Implementation and Assessment of a Life-style Focused Patient Support Application in Myocardial Infarction Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Record Dates: First submitted 2017-06-14; First posted 2017-08-24 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Myocardial Infarction
Keywords: cardiac rehabilitation; eHealth; smartphone application
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (n=50) (No Intervention): Patients randomized to the control arm will receive usual cardiac rehabilitation care post-myocardial infarction.
- Intervention arm: LifePod arm (n=100) (Experimental): In addition to usual cardiac rehabilitation care, patients randomized to the LifePod arm will receive access to the LifePod® support software for six months.
  Interventions: Other: LifePod®

INTERVENTIONS:
Other: LifePod® — The software is a web-based application designed to support persons adhering to lifestyle advice and medication. The patient can log information about lifestyle (i.e. diet, exercise, and smoking), measurements (i.e. weight, pulse and blood pressure), symptoms and medication and can review data in graphs displaying registered values in relation to recommended targets. The software provides positive feedback on healthy choices and gives general recommendations on exercise training, physical activity and healthy diet. Reminders are generated in the case of decreasing registrations. Finally, short text messages (SMS) will be sent out 2-3 times a week with tips on healthy lifestyle.
  Arms: Intervention arm: LifePod arm (n=100)

SUMMARY:
The study will assess the efficacy of a web-based application as a complement to traditional exercise-based cardiac rehabilitation for improvement of secondary prevention outcomes in post-myocardial infarction patients, compared with usual care. The hypothesis is that the intervention enhances patient adherence to lifestyle advice (exercise training, daily physical activity, healthy diet and tobacco abstinence) and medication, resulting in better risk factor control and prognosis as well as increased self-rated health.

DETAILED DESCRIPTION:
It is well documented that participation in cardiac rehabilitation (CR) programs improves risk factor control and therapy adherence, enhances quality of life and reduces recurrent events. However, the current incomplete fulfilment of guideline recommended CR targets is a matter of concern. Also, while international recommendations advocate program flexibility and individual tailoring, most of the current CR programs are rigid, time-limited and demand substantial health care resources. Therefore, all main international heart associations have claimed for the reengineering of CR to enhance access, adherence, and effectiveness. The general call is for the development of innovative and cost-effective CR programs oriented to modify lifestyle and behaviour with sustainable results and that may be easily integrated in the pre-existing health care structures.eHealth i.e. the use of electronic communication and information technologies in health care, offers a whole new array of possibilities to provide clinical care. These include for example distance monitoring via telecommunication and sensors, interactive computer programs and smart phone applications. While there are thousands of available eHealth applications on the market, only a small minority have been tested in a controlled manner with proper guidance from health care personnel. The study will assess the efficacy of a web-based patient support application as a complement to traditional exercise-based CR for improvement of secondary prevention outcomes in post-MI patients, compared with usual care. The hypothesis is that the intervention enhances patient adherence to lifestyle advice (exercise training, daily physical activity, healthy diet and tobacco abstinence) and medication, resulting in better risk factor control and prognosis as well as increased self-rated health. A secondary hypothesis is that complementing the application with an activity tracker (accelerometer in a smart bracelet) will enhance the effect of the intervention.

ELIGIBILITY:
Inclusion criteria

* Age < 75 years. This cut-off is set as only those < 75 years of age are followed in the national Secondary Prevention after Heart Intensive Care Admission (SEPHIA) registry
* Has suffered an MI within the last 2 weeks
* Owns a smartphone and/or has access to internet via a computer or surf pad and can handle the software

Exclusion criteria

* Expected survival < 1 year
* Dementia, severe psychiatric illness or drug abuse
* Severe physical handicap limiting the patient´s ability to participate in exercise-based CR
* Not able to speak or understand the Swedish language
* Three-vessel disease requiring coronary artery bypass grafting

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Change in submaximal exercise capacity in watts (W) | Change between first (2-4 weeks post-MI) and second (4-6 months post-MI) submaximal exercise test conducted at physiotherapist visits
  Submaximal exercise capacity reflects the patients´ level of physical fitness.The submaximal exercise test is performed on a bicycle ergometer according to the World Health Organisation (WHO) protocol, with an increased workload of 25W every 4.5 minutes The initial starting load, 25W or 50W, is decided, based on the patient's exertion history. After two and four minutes of each workload; heart rate, rate of perceived exertion according to Borg's rating of perceived exertion scale (RPE) and subjective symptoms, including chest pain and dyspnea according to Borg's Category Ratio Scale, CR-10, scale are rated. After three minutes, the systolic blood pressure is registered. The exercise test is discontinued at Borg RPE 17 and/or dyspnea 7 on Borg's CR-10 scale.

SECONDARY OUTCOMES:
Change in self-reported health | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Self-reported Health is measured using the Visual Analogue Scale (0-100)
Change in healthy diet index | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  The healthy diet index is a four-item questionnaire used to evaluate dietary habits within the Swedish Secondary Prevention after Heart Intensive Care Admission (SEPHIA) registry
Smoking habits | First (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Whether the patient is a non-smoker, prior smoker or current smoker (self-report)
Change in weight | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Weight measured in kg
Change in BMI | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Weight in kilograms (kg) divided by height in meters (m) square
Change in waist circumference | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Waist circumference measured in cm
Change in systolic blood pressure | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Systolic blood pressure measured after 5 minutes of rest in supine position (mmHg)
Change in diastolic blood pressure | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Diastolic blood pressure measured after 5 minutes of rest in supine position (mmHg)
Change in total cholesterol | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Fasting plasma total cholesterol
Change in LDL cholesterol | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Fasting plasma LDL cholesterol (mmol/L)
Change in HDL cholesterol | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Fasting plasma HDL cholesterol (mmol/L)
Change in triglycerides | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Fasting plasma triglycerides (mmol/L)
Change in fasting plasma glucose | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Fasting plasma glucose (mg/dL)
Change in hemoglobin A1c | Change between baseline, first (6-8 weeks post-MI) and second (12-14 months post-MI) nurse visits post-MI
  Whole-blood hemoglobin A1c (mmol/mol) by International Federation of Clinical Chemistry (IFCC) standards
Changes in self-reported physical activity | Change between baseline, first (2-4 weeks post-MI) and second (4-6 months post-MI) physiotherapist visits post-MI
  Self-reported physical activity, as measured by Haskell and Frändin & Grimby
Uptake | Six months
  The proportion of patients who log on to the patient interface at least once
Adherence | Six months
  The proportion of patients registering data at least twice per week on a weekly basis throughout the intervention period
Number of contacts with the CR staff | 12-14 months
  Number of telephone and physical contacts with the CR staff during the follow-up period
Incident cardiovascular events at one year | One year
  Incidence of cardiovascular events at one year after the index event: hospitalization for a new MI, heart failure or stroke and cardiovascular death
Incident cardiovascular events at three years | Three years
  Incidence of cardiovascular events at three years after the index event: hospitalization for a new MI, heart failure or stroke and cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Margret Leosdottir, MD, PhD, Principal Investigator — Skane University Hospital and Lund University, Malmo, Sweden
Locations (3):
- Sweden (3):
  - Dept of Cardiology, Skane University Hospital, Lund
  - Dept of Cardiology, Skane University Hospital, Malmo
  - Dept of Cardiology, Umeå

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ogmundsdottir Michelsen H, Sjolin I, Back M, Gonzalez Garcia M, Olsson A, Sandberg C, Schiopu A, Leosdottir M. Effect of a Lifestyle-Focused Web-Based Application on Risk Factor Management in Patients Who Have Had a Myocardial Infarction: Randomized Controlled Trial. J Med Internet Res. 2022 Mar 31;24(3):e25224. doi: 10.2196/25224. PMID 35357316
- [Derived] Gonzalez M, Sjolin I, Back M, Ogmundsdottir Michelsen H, Tanha T, Sandberg C, Schiopu A, Leosdottir M. Effect of a lifestyle-focused electronic patient support application for improving risk factor management, self-rated health, and prognosis in post-myocardial infarction patients: study protocol for a multi-center randomized controlled trial. Trials. 2019 Jan 24;20(1):76. doi: 10.1186/s13063-018-3118-1. PMID 30678709
- See also: Cross Technology Solutions home page — http://www.cross-solutions.com/